CLINICAL TRIAL: NCT01361282
Title: Evaluation of Total Corneal Power Calculations for Intraocular Lens Selection Using the Optovue OCT in Descemet's Stripping Automated Endothelial Keratoplasty (DSAEK) Patients
Brief Title: Using the Optovue OCT to Select IOL Power
Status: Terminated | Type: Observational
Why Stopped: The DSAEK procedure was discontinued as the standard of care for the intended cohort.
Sponsor: Legacy Health System (Other)
Collaborators: Devers Eye Institute (Other); Optovue (Industry); Lions VisionGift Research (Other)
Responsible Party: Principal Investigator, Mark A Terry, Director of Corneal Services, Legacy Health System
Other Study IDs: LEBO-2011-1
Record Dates: First submitted 2011-05-25; First posted 2011-05-26 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Fuchs' Endothelial Dystrophy; Cataract
Keywords: Total Corneal Power; Optical Coherence Tomography; Descemet Stripping Endothelial Keratoplasty
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Triple Procedure: All qualifying patients will have received DSAEK with concurrent cataract extraction and intraocular lens placement. Data collection will occur between 6-18 months post-operation.

SUMMARY:
Many patients with endothelial dysfunction also present with cataracts. It is therefore common practice to perform cataract extraction and intraocular lens (IOL) implantation during the same operation and immediately prior to Descemet's Stripping Automated Endothelial Keratoplasty (DSAEK), in order to minimize trips to the operating room and the associated risks of ocular surgery. However, the unique posterior corneal anatomy of the DSAEK recipient makes it difficult to predict pre-operatively the proper power of IOL to place, and some patients end up with a mismatched lens that requires spectacle correction. The current gold standard for IOL power calculation (A-Scan optical biometry) takes measurements of the anterior surface of the cornea and makes assumptions about the posterior surface that are violated by the unique hourglass shape of the donor DSAEK graft. New optical coherence tomography (OCT) technology provides us with the ability to measure curvature in both the anterior and posterior aspects of the cornea in order to generate an IOL calculation that has the potential to give more accurate results for our DSAEK patients.

The investigators will be using the Optovue to perform corneal power analysis on patients who have already received DSAEK and cataract surgery, in order to compare the post-op Optovue power calculations to the pre-operative power calculations provided by the A-Scan. If the OCT is shown to provide accurate IOL power calculations, then some patients might be better served by a two-stage procedure where DSAEK is performed and then followed six months later by cataract surgery using the OCT to calculate IOL power.

ELIGIBILITY:
Inclusion Criteria:

* 18 year of age or older
* Diagnosis of Fuchs' Endothelial Dystrophy with cataract
* Recent history of DSAEK with concurrent phacoemulsification & intraocular lens (IOL) implantation

Exclusion Criteria:

* Diagnosis of ocular comorbidity that might be limiting to visual acuity (glaucoma, retinal disease, surface irregularities, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All study subjects will have received Descemet's Stripping Automated Endothelial Keratoplasty (DSAEK) for Fuchs' Endothelial Dystrophy, together with concurrent cataract surgery. Data collection will occur between 6 and 18 months following surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-11-09 (Actual); Primary Completion 2016-09-09 (Actual); Study Completion 2016-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Terry, MD, Principal Investigator — Devers Eye Institute
Locations (1):
- Devers Eye Institute, Portland, Oregon, United States